CLINICAL TRIAL: NCT06370481
Title: HIV, Equity, and Addiction Training (HEAT) Program
Acronym: HEAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ellen Eaton, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012349; K24DA060786 (NIH)
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorders; Hiv; Opioid Use Disorder; Stimulant Use (Diagnosis)
Keywords: Alabama; Ryan White Clinics; HIV treatment; Substance use disorder treatment; Telemedicine
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Disease | interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients living with HIV and substance use (Experimental): Patients living with HIV and substance use, aged 18 and over. These participants are receiving services at HIV clinics in Alabama and must have reported opioid and/or stimulant misuse.
  Interventions: Other: Telemedicine; Other: Standard of care

INTERVENTIONS:
Other: Telemedicine — Routine care administered via telemedicine
Other: Standard of care — Standard of care, as received in HIV clinic settings

SUMMARY:
This project is a pilot study to determine the feasibility and acceptability of a telemedicine intervention for substance use disorder service delivery in diverse people living with HIV in Alabama.

DETAILED DESCRIPTION:
The contemporary drug crisis and the COVID-19 pandemic have exposed the complex syndemics of addiction and infectious diseases: rising rates of substance use disorder (SUD) have outpaced our ability to respond with a limited healthcare workforce and public health capacity. SUD is increasing in those living with and at risk for HIV, and infectious consequences of SUD, like hepatitis C, have continued, unmitigated, in rural parts of the U.S. where many states lack Medicaid expansion, syringe service programs, and public health infrastructure to respond to the drug crisis and comorbid infections. Systemic racism and regressive policies in the Deep South criminalize people who use drugs, creating additional barriers to care, HIV prevention, and addiction treatment. As a result, people who use drugs rarely receive comprehensive addiction and HIV treatment. Yet telemedicine has the potential to overcome these barriers and bypass the constraints of a brick-and-mortar clinic to link vulnerable people, including those with HIV, to care. Although telemedicine has become mainstream in recent years, few studies have evaluated telemedicine for SUD in the Deep South from the perspective of patients and providers.

ELIGIBILITY:
Inclusion Criteria:

* Receiving services at HIV clinics in Alabama
* Reported opioid and/or stimulant misuse
* 18 years of age or older

Exclusion Criteria:

* Receipt of SUD clinical care other than through HIV provider/clinic in the last 3 months
* Inability to engage in interviews independently without support (e.g., cognitive impairment)
* Currently psychotic
* Actively suicidal: presents with a suicide attempt or suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — At least 20% female, no more than 80% male
Enrollment: 30 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who have a follow-up healthcare visit | 1 month, 2 months, 3 months
  Follow up visit for care (either telemedicine or in person)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen F Eaton, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The research will comply with the NIH Data Sharing policy and will coordinate collection and sharing of key data. Data are available upon request from the public and research community after main findings are published. To request data, the investigators ask that interested parties submit a detailed description of the aims and methods of their research to the PI, including contact information from the primary requester, institutional affiliation, current CV and qualifications, sources of financial support, and conflict of interest statement. The MPIs will review requests as submitted and determine the appropriateness of the request with collaborators or if additional safeguards are needed. Upon approval, data transfer agreements must be established and proof of IRB approval from the requester's institutional IRB must be presented. Our team will comply with HIPAA and Common Rule de-identification prior to data sharing to ensure protection of study participants
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available after studies are published and will be maintained for 5 years after study end date.